CLINICAL TRIAL: NCT02549079
Title: Soluble Factors in the Serum of Severely Burned Patients
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: EK104/08
Record Dates: First submitted 2015-09-11; First posted 2015-09-14 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Burn Patients
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Blood sample — Blood will be taken from all patients meeting the inclusion criteria.

SUMMARY:
The present study investigates the levels of certain soluble factors in the blood of patients with severe burn injury. Serum levels of different soluble factors will be correlated with the clinical outcome, presence of sepsis, the area of burn, and other clinical parameters in order to make a statement regarding their use as biomarkers in the prediction and monitoring of burn patients.

DETAILED DESCRIPTION:
Burn patients still represent a critical patient collective with a high mortality rate although treatment technologies have improved over the years. One problem healthcare professionals face is the fact that reliable biomarker which predict the clinical outcome, the onset of sepsis, and monitor the severity of disease in burn patients are still missing. These biomarkers would allow an early adoption of treatment modalities to improve the outcome and prevent life-threatening complications.

Blood samples from severely burned patients will be collected over a period of five days and different cytokines (for example the macrophage migration inhibitory factor protein family) will be measured in the serum. Clinical data of the patients (sepsis, total body surface area of burns, abbreviated burn severity index, sepsis-related organ failure assessment, etc.) will be documented and correlated to the levels of soluble factors.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* minimum of 10% total body surface area burn
* needing ICU treatment

Exclusion Criteria:

* younger than 18 years of age
* immunosuppression (e.g. HIV)
* undergone surgery 2 weeks prior to burn injury
* malignancies
* severe diseases (myocardial infarction, lung embolism)
* declining to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with burn injuries treated in the burn intensive care unit
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2004-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Survival of a total of 23 burn patients during their treatment in the ICU | five days
  Patients will be monitored over five days and death (with underlying condition, time) will be determined and documented by medical doctors.

SECONDARY OUTCOMES:
Onset of sepsis of a total of 23 burn patients during their treatment in the ICU | five days
  Onset of systemic inflammatory response syndrome, sepsis, septic shock will be monitored by medical doctors by standardized assessment of clinical parameters according to the consensus of the American College of Chest Physicians (ACCP) and the Society of Critical Care Medicine (SCCM) (released in Critical Care Med, 20(6):864-74, 1992, Pubmed ID: 1597042)

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Pallua, M.D., Ph.D., Principal Investigator — RWTH Aachen University